CLINICAL TRIAL: NCT04329637
Title: An Integrative, Patient-Centered Model of Care: Meditation and Care Coordination to Improve Healthcare Outcomes in Cyclic Vomiting Syndrome
Brief Title: Effects of an Integrative Health Care Model With Meditation and Care Cordination in CVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Thangam Venkatesan, Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00027409
Record Dates: First submitted 2020-03-26; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Cyclic Vomiting Syndrome
Keywords: cyclic vomiting; meditation; care coordination
MeSH Terms: conditions — Familial cyclic vomiting syndrome

STUDY DESIGN:
Intervention Model Description: Patients were prospectively randomized to either the integrative health care model (IHC model) or usual care (UC)/control group after signing informed consent. Demographics, clinical characteristics and outcomes of interest were measured at baseline before the intervention, and at 3 and 6 months. Global psychological distress ,depression, catastrophizing, anxiety/pain-related fear, and social support were assessed using validated tools. Coping skills were measured with the validated short version of the COPE questionnaire. Quality of sleep was assessed using Pittsburgh Sleep Quality Index (PSQI). HRQoL was measured with the NIH PROMIS Short Forms. Health care utilization was recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IHC (intergrative health care) arm (Active Comparator): Meditation and care coordination in addition to usual care
  Interventions: Other: Integrative healt care
- usual care (No Intervention): usual care

INTERVENTIONS:
Other: Integrative healt care — Meditation and use of a care cordinator
  Other Names: IHC
  Arms: IHC (intergrative health care) arm

SUMMARY:
Cyclic vomiting syndrome is a chronic functional gastrointestinal disorder that is a significant health care problem. It affects 1-2% of the population and imposes an enormous burden on patients, families and the health care system. Due to the recalcitrant nature of the disease, patients have high rates of health care utilization with multiple emergency department visits and hospitalizations. These in turn lead to school and work absenteeism, job loss, divorce and even disability. CVS is also associated with multiple comorbid conditions such as anxiety and depression, which further contribute to disease severity. Both neuroimaging studies and other data demonstrate the role of the central nervous system in the pathophysiology of CVS with stress being a significant trigger for episodes of CVS. In summary, CVS is common, disabling and expensive and is associated with significant psychosocial comorbidity that contributes to impaired quality of life . Our current healthcare delivery model is disease-centric and does not adequately address the psychosocial barriers that contribute to poor health in this patient population. We propose a novel, collaborative, integrative health care model that shifts the paradigm of care from one that is episodic and disease-centered to a patient-centered approach that addresses psychosocial determinants of health not addressed in our current traditional health care system. We will incorporate meditation practices that have been shown to reduce psychological distress and also add a care coordinator to our health care delivery team. The primary role of the care coordinator is to identify patient goals, preferences and barriers to self-management and address psychosocial and environmental issues that determine health. Patients will be randomized to either the integrative health care model or usual care. The primary aim of our study is to determine the impact of our proposed integrative health care model on health care outcomes which will include a reduction in psychological distress, improvement in coping skills for managing chronic disease, cognitive symptom management, improvement in health-related quality of life and reduction in health care utilization. This collaborative effort between physicians, community partners, and allied health personnel will redesign the health care delivery system, facilitate access to appropriate healthcare services, optimize chronic disease management and improve overall healthcare outcomes.

DETAILED DESCRIPTION:
Background & Aims: Cyclic vomiting syndrome (CVS) is associated with psychosocial comorbidity and often triggered by stress. The current disease-centered model of care does not address psychosocial factors that impact patient outcomes. The investigators hypothesized that a holistic, patient-centered care model integrating meditation and addressing psychosocial needs through a care coordinator, will improve healthcare outcomes in CVS.

Methods: The investigators conducted a prospective randomized controlled trial of 49 patients with CVS (mean age: 34 ± 14 years; 81% female) who were randomized to conventional healthcare (control group) or Integrative Health Care (IHC) (27: control group, 22: IHC group;). In the IHC group, patients were assigned a care coordinator and received meditation sessions from certified trainers from the Heartfulness Institute. Outcomes including psychological distress, coping strategies to manage chronic stress, cognitive symptom management, and Health-Related Quality of Life were measured with validated tools. An intention-to-treat analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* All subjects with CVS

Exclusion Criteria:

* Severe cognitive impairment, active mental health problems such as suicidal ideation, severe anxiety or depression requiring inpatient care, or an inability to sit for at least 20 minutes. Subjects with severe cardiopulmonary diseases, malignancy, liver cirrhosis, renal failure on dialysis or those who were pregnant at the time of enrollment were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Levels of psychological distress is measured using a validated questionnaire called the Basic Symptom Inventory | 6 months
  Basic symptom inventory The Brief Symptom Inventory (BSI) consists of 53 items covering nine symptom dimensions: Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism; and three global indices of distress: Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. The global indices measure current or past level of symptomatology, intensity of symptoms, and number of reported symptoms, respectively.

SECONDARY OUTCOMES:
Mutiple domains of coping will be measured by the COPE questionanire which is a validated tool | 6 months
  COPE questionanire: The COPE questionnaire consists of the following. Five scales (of four items each) measure conceptually distinct aspects of problem-focused coping (active coping, planning, suppression of competing activities, restraint coping, seeking of instrumental social support); five scales measure aspects of what might be viewed as emotional-focused coping (seeking of emotional social support, positive reinterpretation, acceptance, denial, turning to religion); and three scales measure coping responses that arguably are less useful (focus on and venting of emotions, behavioral disengagement, mental disengagement).

IPD SHARING:
Plan to Share IPD: No